CLINICAL TRIAL: NCT03454373
Title: Long Term Follow-Up of Food and Cash Assistance for HIV-Positive Men and Women on Antiretroviral Therapy in Tanzania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Ministry of Health and Social Welfare, Tanzania (Other Government)
Responsible Party: Principal Investigator, Sandra McCoy, Assistant Adjunct Professor, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-11-10508
Record Dates: First submitted 2018-02-15; First posted 2018-03-05 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Hiv
Keywords: HIV; Food Insecurities; Antiretroviral Therapy
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentive for return to care (Experimental): Standard of care HIV primary care services, including counseling to return to care, plus a one-time "re-start" incentive of 22,500 TZS to return to care.
  Interventions: Behavioral: Incentive for linkage to care
- Comparator (No Intervention): Standard of care HIV primary care services, including counseling to return to care.

INTERVENTIONS:
Behavioral: Incentive for linkage to care — Participants who were found to have been lost to care will receive standard of care plus a one-time "re-start" incentive of 22,500 TZS to return to care
  Arms: Incentive for return to care

SUMMARY:
This protocol is for the long term follow-up study of "Comparing Food and Cash Assistance for HIV-Positive Men and Women on Antiretroviral Therapy (ART) in Tanzania", a 3-arm randomized controlled trial led by Professor Sandra McCoy at the University of California Berkeley and Dr. Prosper Njau at the Tanzanian Ministry of Health and Social Welfare. The investigators will determine the long-term effectiveness of short-term incentives for ART adherence and retention in care. The study will also determine whether incentives can also be used to re-engage PLHIV with HIV care after they have fallen out of care.

DETAILED DESCRIPTION:
This study will build on preliminary data from a randomized study conducted in Shinyanga, Tanzania which found that short-term cash and food assistance improved ART adherence and retention in care among food insecure people living with HIV infection (PLHIV) after 6 and 12 months of follow-up. The investigators will now determine the long-term effectiveness of these incentive strategies. In this 2-year study, investigators will first determine 24-month adherence and retention outcomes using medical and pharmacy records for the 781 PLHIV who were alive at the end of the previous study, which concluded after 12 months of follow-up (Aim 1). Then, leveraging an existing program of home based care, investigators will determine the prevalence of undocumented transfers and deaths among the subset of patients found to be lost to follow-up or transferred in clinic records. Investigators will use these data from home visits to adjust estimates of the interventions' effectiveness on retention in HIV care and mortality (Aim 2). Among the PLHIV found to be disengaged from care, investigators will conduct a pilot study of a one-time cash incentive to encourage PLHIV to re-engage with care, with the goal of mitigating the barriers posed by transportation and opportunity costs (Aim 3). At the conclusion of the project, investigators will understand the long-term effectiveness of cash and food incentives for adherence and retention, and whether they can also be used for re-linking PLHIV to care, data highly relevant to 'Treat All' programs in Fast Track countries.

ELIGIBILITY:
Inclusion Criteria:

* Study participant in the prior study "Comparing Food and Cash Assistance for HIV-Positive Men and Women on Antiretroviral Therapy in Tanzania" (NCT01957917)
* Alive and willing to provide written informed consent
* Not currently enrolled in HIV care services

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
The proportion of PLHIV linked to HIV care at 3 months | 3 months
  Initial re-engagement in care, defined as as the proportion of PLHIV who have completed (attended) a HIV primary care visit at the clinic of the PLHIV's choosing within 3 months of the incentive offer to return to care.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra I McCoy, MPH, PhD, Principal Investigator — University of California, Berkeley
Locations (3):
- Tanzania (3):
  - Kambarage Health Center, Shinyanga, Shinyanga
  - Shinyanga Regional Hospital, Shinyanga, Shinyanga
  - Kahama District Hospital, Shinyanga